CLINICAL TRIAL: NCT02835365
Title: Observational Study on Patients With Baclofen Treatment for Alcohol-dependence in French Gastro and Hepatology Departments
Brief Title: Observational Study on Patients With Baclofen Treatment for Alcohol-dependence in France
Acronym: OBADE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Principal Investigator, Camille Barrault, Dr, Centre Hospitalier Intercommunal Creteil
Other Study IDs: OBADE
Record Dates: First submitted 2016-07-11; First posted 2016-07-18 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Alcohol Drinking; Cirrhosis; Alcohol Withdrawal
Keywords: baclofen; alcohol; withdrawal
MeSH Terms: conditions — Alcohol Drinking; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — biologic sample to dose the blood baclofenemia
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients treated with baclofen: Patients treated with baclofen to diminish their alcohol consumption in the ANGH centers will be enrolled

SUMMARY:
Baclofen is an agonist of the amino-butyricum B (GABA-B) receptor used for a long time in neurology to treat spastic contracture. Several clinical studies have suggested its efficacy in the treatment of alcohol-dependence in low, even in case of cirrhosis and high dose. French drug authority has authorized its use in 2012 whereas the l'European Association for the Study of the Liver recommends to perform additional studies on this indication.

The goal of this observational study is to evaluate the use of baclofen for alcohol-dependence in real life care as well its efficacy.

DETAILED DESCRIPTION:
Numerous centers of the French research group of the national association of the hepatologists and gastroenterologists from general hospitals (ANGH) will be part of this study. Patients treated with baclofen for alcohol -dependence will be enroll prospectively from 2014 and retrospectively if they were treated between 2012 and 2014. The reported alcohol consumption, biological markers of excessive alcohol, initial and usual baclofen dosage, blood balofen dosage as well as clinical data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years old
* patient treated with baclofen therapy after 2012 for alcoholo-dependance

Exclusion Criteria:

* Baclofen therapy before 2012
* patient who refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients older than 18 years old and who received a baclofen therapy for alcohol-dependance after 2012 in a participating site is eligible. The referral physician must inform the patient. Only patients who give their oralm accceptance will be included.
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Target population | at inclusion
  Demographic and clinical characteristics of patients who take baclofen for alcohol addiction: mean age, alcohol consumption, child pugh score, etc.

SECONDARY OUTCOMES:
baclofen posology | at inclusion, at 3, 6 and 12 months of follow-up
  used baclofen posology will be recorded to determine the posology scheme to treat patients with or without cirrhosis
Alcohol consumption | at inclusion, at 3, 6 and 12 months of follow-up
  Evolution of the alcohol consumption in patients under baclofen therapy
Biological markers of alcohol consumption | at inclusion, at 3, 6 and 12 months of follow-up
  Evolution of the biological markers of alcohol consumption in patients under baclofen therapy
baclofen tolerance | at 3, 6 and 12 months of follow-up
  Description of the side effects under baclofen therapy
Baclofen dosage | at 3, 6 and 12 months of follow-up
  Blood baclofen dosage under baclofen treatment, if available

CONTACTS AND LOCATIONS:
Overall Officials: Camille barrault, MD, Principal Investigator — CHI Créteil
Locations (8):
- France (8):
  - Centre hospitalier yves LEFOLL, Saint-Brieuc, Côtes d'Armor
  - Centre Hospitalier Régional Universitaire Hôpital Jean Minjoz, Besançon, Franche-Comté
  - CH Béziers, Béziers, Hérault
  - CH Orleans, Orléans, Loiret
  - GHPSO Creil-Senlis, Creil, Oise
  - CH meaux, Meaux, Seine Et Marne
  - CHI CRETEIL addictology, Créteil
  - Hôpital saint denis, Saint-Denis, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No